CLINICAL TRIAL: NCT03211897
Title: Prospective Observational Investigation of Olanzapine Versus Haloperidol Versus Ziprasidone Versus Midazolam for the Treatment of Acute Undifferentiated Agitation in the Emergency Department
Brief Title: Olanzapine, Haloperidol, Ziprasidone, Midazolam for Acute Undifferentiated Agitation
Acronym: MOHZA
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HSR # 17-4345
Record Dates: First submitted 2017-06-26; First posted 2017-07-07 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Agitation,Psychomotor
MeSH Terms: conditions — Psychomotor Agitation | interventions — Haloperidol; ziprasidone; Olanzapine; Midazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Haloperidol 5mg Intramuscular: As part of the quality initiative protocol, patients who are treated for acute agitation in the ED will receive haloperidol as their initial sedative agent during the 21 day block. All subsequent agitation medications are at the discretion of the provider.
  Interventions: Drug: Haloperidol Injection
- Ziprasidone 20mg Intramuscular: As part of the quality initiative protocol, patients who are treated for acute agitation in the ED will receive ziprasidone as their initial sedative agent during the 21 day block. All subsequent agitation medications are at the discretion of the provider.
  Interventions: Drug: Ziprasidone Injection
- Olanzapine 10mg Intramuscular: As part of the quality initiative protocol, patients who are treated for acute agitation in the ED will receive olanzapine as their initial sedative agent during the 21 day block. All subsequent agitation medications are at the discretion of the provider.
  Interventions: Drug: OLANZapine Injection
- Midazolam 5mg Intramuscular: As part of the quality initiative protocol, patients who are treated for acute agitation in the ED will receive midazolam as their initial sedative agent during the 21 day block. All subsequent agitation medications are at the discretion of the provider.
  Interventions: Drug: Midazolam injection

INTERVENTIONS:
Drug: Haloperidol Injection — As part of the quality initiative protocol, patients who are treated for acute agitation in the ED will receive haloperidol as their initial sedative agent during the 21 day block. All subsequent agitation medications are at the discretion of the provider.
  Groups: Haloperidol 5mg Intramuscular
Drug: Ziprasidone Injection — As part of the quality initiative protocol, patients who are treated for acute agitation in the ED will receive ziprasidone as their initial sedative agent during the 21 day block. All subsequent agitation medications are at the discretion of the provider.
  Groups: Ziprasidone 20mg Intramuscular
Drug: OLANZapine Injection — As part of the quality initiative protocol, patients who are treated for acute agitation in the ED will receive olanzapine as their initial sedative agent during the 21 day block. All subsequent agitation medications are at the discretion of the provider.
  Groups: Olanzapine 10mg Intramuscular
Drug: Midazolam injection — As part of the quality initiative protocol, patients who are treated for acute agitation in the ED will receive midazolam as their initial sedative agent during the 21 day block. All subsequent agitation medications are at the discretion of the provider.
  Groups: Midazolam 5mg Intramuscular

SUMMARY:
The goal of this research investigation is to conduct a prospective observational study of the comparative efficacy of haloperidol versus olanzapine versus midazolam versus ziprasidone for the treatment of acute undifferentiated agitation in the emergency department.

DETAILED DESCRIPTION:
The ED will implement a treatment protocol as a quality improvement initiative. All patients requiring chemical sedation for will receive haloperidol as the initial treatment for agitation for 21 days, followed by ziprasidone as the initial treatment for agitation for 21 days, followed by olanzapine as the initial treatment for agitation for 21 days, and finally midazolam as the initial treatment for agitation for 21 days.

This is a clinical care quality improvement protocol. The research component is the observation of this clinical care protocol.

Patients who receive medications in the ED will be observed by research staff, evaluating efficacy and safety of the administered medication. The decision to administer the medication is at the discretion of the physician. Research protocols are only such that we are observing the efficacy and safety, which coincides the quality improvement purposes of this clinical protocol.

Trained Research Associates will collect all data on patients who receive a protocol medication. This will include baseline demographic data including age, gender, etiology of agitation (according to the treating physician, presumed at the time of medication administration), initial vital signs, breath alcohol level, drug screen results, pre-hospital medications administered, and any other laboratory data available at the time (e.g. glucose).

Research associates will record the patient's level of agitation using a validated agitation scale, the Altered Mental Status (AMS scale). The AMS scale is an ordinal scale ranging from -4 (profoundly somnolent) to +4 (profoundly agitated), with agitation generally defined as an AMS scale of 2 or greater. This scale is a modified version of the Observer's Assessment of Alertness Scale and the Behavioral Activity Rating Scale.

AMS scores will be recorded at the time of medication administration and at every subsequent 15-minute interval until 120 minutes. Research associates will also carry stopwatches and record the time elapsed until adequate sedation (defined as an AMS ≤ 0), as well as whether other medications (defined as "rescue medications") were administrated for any reason and at what time this occurred.

Research associates will prospectively monitor each patient for all adverse side effects of the medications, including hypoxia, need for airway intervention (nasal cannula, facemask, non-invasive positive pressure ventilation, endotracheal intubation), hypotension, cardiac dysrhythmias, extrapyramidal side effects, and other complications.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department patients (18+) with acute undifferentiated agitation requiring chemical sedation at the discretion of the attending emergency physician

Exclusion Criteria:

* Known pregnancy
* Allergy to the medication during the block
* Prisoner/under arrest

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Emergency Department patients with acute undifferentiated agitation requiring chemical sedation at the discretion of the attending emergency physician. Patients studied are from a population where agitation is predominantly due to alcohol, illicit substances, or psychiatric agitation.
Sampling Method: Probability Sample
Enrollment: 737 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the mean difference in Altered Mental Status (AMS) score from baseline at 15 minutes post-administration for each study drugs. | 15 minutes
  Patients score on a previously validated agitation scale called the AMSS
  ADDENDUM: The primary outcome for this study was changed prior to study initiation to the proportion of patients adequately sedated at 15 minutes (defined as AMSS < 1). This addendum was methodologically necessary to account for the ordinal, non-normal distribution of this data.

SECONDARY OUTCOMES:
Time to adequate sedation | Within the 120 minutes post-medication administration
  The time elapsed in minutes to achieve a score of < 1 on a validated agitation scale called the AMSS
Rescue Sedation | 1 hour
  Proportion of patients requiring additional medication for sedation within 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Klein, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klein LR, Driver BE, Miner JR, Martel ML, Hessel M, Collins JD, Horton GB, Fagerstrom E, Satpathy R, Cole JB. Intramuscular Midazolam, Olanzapine, Ziprasidone, or Haloperidol for Treating Acute Agitation in the Emergency Department. Ann Emerg Med. 2018 Oct;72(4):374-385. doi: 10.1016/j.annemergmed.2018.04.027. Epub 2018 Jun 7. PMID 29885904